CLINICAL TRIAL: NCT04404205
Title: The Effect of Cochlear Implant on Postural Control
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Chief of Department Otolaryngology, Pamukkale University
Other Study IDs: 6
Record Dates: First submitted 2020-05-17; First posted 2020-05-27 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Cochlear Implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patient with cochlear implant: Adult patients who had cochlear implant surgery before will be included. We will call patients from our cochlear implant list.
  Interventions: Diagnostic Test: Postural stability measurements by Biodex Balance System

INTERVENTIONS:
Diagnostic Test: Postural stability measurements by Biodex Balance System — Postural stability measurements will be done by Biodex Balance System. Three preprogrammed main tests will be applied. Postural stability, fall index, sensory integration will be calculated. All tests will be done in four conditions; implant off(1), implant on(2), implant on music on(3), and implant off again(4).

SUMMARY:
Some patients are having balance problems after cochlear implant surgery. There are contradictory reports about the effect of the implant on postural control. While the cochlear implant is working, an electrical current is continuously stimulating the cochlear nerve which is in close proximity with vestibular ganglion and nerve. This stimulation may contribute to vestibular signals to the central system. The aim of the study is to investigate if this stimulation has any effect on postural control.

DETAILED DESCRIPTION:
Adult patients who had unilateral cochlear implantation will be included. Postural stability measurements will be done by the Biodex Balance System. Three preprogrammed main tests and their 9 subtests will be applied. Postural stability, fall index, sensory integration will be calculated. All tests will be done in four conditions; implant off(1), implant on(2), implant on music on(3), and implant off again(4).

ELIGIBILITY:
Inclusion Criteria:

* Patients who had cochlear implant surgery before

Exclusion Criteria:

* Bilateral Cochlear implants
* Neurologic disease
* Communication problem
* Additional disability

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had cochlear implantation in our hospital will be invited to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Deviation of center of gravity(angle) | 3-6 months
  Deviation of center of gravity(angle) test assesses a patient's ability to maintain a center of balance. It measures how much the patient's position deviates from center and reports the average deviation as the stability index. Therefore, a low score is more desirable than a high score. Postural stability is a calculated value of difference in center of gravity when the subjects tested eyes open/closed, hard and soft surface test conditions. Postural stability will be measured in four conditions: İmplant on, implant off, implant on+music on, implant of again
postural sway velocity(angle/sec) | 3-6 months
  A high sway velocity when a patient is attempting to stand motionless suggests a deficit in postural control and assessment for lower extremity strength, proprioception, and vestibular or visual deficiencies. Postural sway velocity will be measured in four conditions: İmplant on, implant off, implant on+music on, implant of again
Sensory Integration Test(the mean absolute deviation of the patient's average position during a test) | 3-6 months
  The Clinical Test of Sensory Interaction of Balance (CTSIB) is a standard test for balance assessment on a static surface. The test assesses how well a patient can integrate sensory information to maintain balance. The result of the CTSIB test is the patient's sway index, which represents the mean absolute deviation of the patient's average position during a test. The higher the sway index, the more unsteady the person was during the test. Sensory Integration Test will be measured in four conditions: İmplant on, implant off, implant on+music on, implant of again

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl N Ardıç, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be available University depository